CLINICAL TRIAL: NCT02480842
Title: Randomized Clinical Trial With Two Physical Therapy Protocols After Breast Cancer Surgery and Immediate Reconstruction
Brief Title: Clinical Trial With Two Physical Therapy Protocols After Breast Cancer Surgery and Immediate Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, FUSaoPaulo PT3, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSaoPaulo PT 3
Record Dates: First submitted 2015-06-17; First posted 2015-06-25 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Mammaplasty; Breast Implantation; Range of Motion, Articular; Shoulder Joint; Physical Therapy Modalities
MeSH Terms: conditions — Breast Neoplasms

ARMS (4):
- Alloplastic group A (Experimental): After randomization (15 days after surgery):
  - Patients will start to perform exercises with free shoulder ROM. Patients will be told only to limit the movement if they feel pain.
  Interventions: Other: Alloplastic free ROM
- Alloplastic group B (Experimental): After randomization (15 days after surgery):
  - Patients will keep shoulder exercises limited to 90° up to 30 days after surgery. At that moment (one month after surgery), then patients will also be allowed to move the shoulder with no restriction
  Interventions: Other: Alloplastic limited ROM
- Oncoplastic group A (Experimental): After randomization (15 days after surgery):
  - Patients will start to perform exercises with free shoulder ROM. Patients will be told only to limit the movement if they feel pain.
  Interventions: Other: Oncoplastic free ROM
- Oncoplastic group B (Experimental): After randomization (15 days after surgery):
  - Patients will keep shoulder exercises limited to 90° up to 30 days after surgery. At that moment (one month after surgery), then patients will also be allowed to move the shoulder with no restriction
  Interventions: Other: Oncoplastic limited ROM

INTERVENTIONS:
Other: Alloplastic free ROM
  Arms: Alloplastic group A
Other: Alloplastic limited ROM
  Arms: Alloplastic group B
Other: Oncoplastic free ROM
  Arms: Oncoplastic group A
Other: Oncoplastic limited ROM
  Arms: Oncoplastic group B

SUMMARY:
Introduction: physical therapy is essential in preventing motor and functional complications after breast cancer surgery. However, there is no prospective randomized study of different physiotherapy approaches in patients undergoing breast cancer surgery with immediate reconstruction. Objectives: to evaluate two physical therapy protocols in patients after breast cancer surgery with immediate reconstruction. A group with shoulder exercises with limited range of motion (ROM) at 90 degrees up to a month after surgery and a group with limited ROM only up to 15 days after surgery. Specific objectives: to evaluate shoulder ROM and pain one week before the surgery on average, and 07, 15, 30, 60, 90 and 180 days after surgery; assess motor function one week before the surgery on average, and 30 and 90 days after surgery; evaluate dehiscence and seroma 07, 15, 30, 60 and 90 days after surgery; associate incidence of seroma and dehiscence with preoperative risk factors and compare all variables (shoulder ROM, pain, motor function, seroma and dehiscence) between the two groups. Methods: women with breast cancer, who will be submitted to breast surgery (radical or conservative), followed by immediate reconstruction: alloplastic (tissue expander or breast implant) or oncoplastic (breast reduction or contralateral symmetrization) will be included. Patients that will be submitted to bilateral oncology surgery, reconstruction with autologous tissue or breast surgery without reconstruction will not be included. Patients will be recruited just after surgery scheduling and will undergo preoperative evaluation. At this moment, preoperative analysis will be conducted with personal data and medical history. Patients will undergo new assessments 07, 15, 30, 60, 90 and 180 days after surgery. All patients will receive standard physiotherapy treatment for women undergoing breast reconstruction from Physical Therapy Sector. The protocol consists of early exercise, limited to 90° of shoulder ROM, starting the day after the surgery and repeated 7 days after surgery. After 15 days of surgery, the patients will be randomized into two treatment protocols. One group will start to perform exercises with free shoulder ROM. Patients will be told only to limit the movement if they feel pain. The other group will keep shoulder exercises limited to 90° up to 30 days after surgery. At that moment (one month after surgery), they will also be allowed to move the shoulder with no restriction. The evaluation of the presence of dehiscence and seroma will occur by inspection and palpation. Shoulder ROM will be investigated through active goniometry of flexion, extension, adduction, abduction, internal rotation and external rotation. The pain will be assessed with the Verbal Numerical Scale from 0 to10 and upper limb function through the DASH (Disabilities of the Arm, Shoulder and Hand Questionnaire) questionnaire.

DETAILED DESCRIPTION:
Methods:

Patients will be recruited just after surgery scheduling. They will undergo preoperative evaluation one week before the surgery on average. At this moment, preoperative analysis will be conducted with personal data and medical history. Patients will undergo new assessments 07, 15, 30, 60, 90 and 180 days after surgery, periods that will be described as PO 07, PO 15, PO 30, PO 60, PO 90 and PO 180.

All patients will receive standard physiotherapy treatment for women undergoing breast reconstruction from Physical Therapy Sector of Mastology Discipline of the Department of Gynecology of Federal University of São Paulo. The protocol consists of early exercise, limited to 90° of shoulder range of motion (ROM), starting the day after the surgery and repeated 7 days after surgery.

After 15 days of surgery, the patients will be randomized into two treatment protocols.

However, because of the existence of different types of reconstructive surgery, randomization will performed from two groups:

* Alloplastic group: patients who will undergo reconstruction with tissue expander or breast implant
* Oncoplastic Group: patients who will undergo mammaplasty and / or contralateral symmetrization

Computer random sequence will be used for randomization, in which each group will be randomized to Group A or Group B.

* Subgroup A: Patients will start to perform exercises with free shoulder ROM. Patients will be told only to limit the movement if they feel pain.
* Subgroup B: Patient will keep shoulder exercises limited to 90° up to 30 days after surgery. At that moment (one month after surgery), then patients will also be allowed to move the shoulder with no restriction

At the end of randomization there will be four subgroups: alloplastic A, alloplastic B, oncoplastic A and oncoplastic B

Outcomes:

1. Shoulder range of motion:

   The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively. The patient will be positioned in the sitting position. To assess shoulder flexion, the upper limb will be in neutral position with elbow extension. Patient will be asked to raise the arm forward, close to the body. To assess extension, the arm will be positioned with 90° of elbow flexion and the patient will be asked to take the arm back. For adduction, the patient will be with 90° of shoulder flexion with the palm down and patient will be told to move the arm medially. For the study of the upper limb abduction, the limb will be in supination and elbow extension and the patient will be asked to raise the arm to the side, along the trunk line toward the ear. For the evaluation of internal rotation and external rotation the upper limb will be placed in 90° of shoulder abduction and 90° of elbow flexion. The patient will be asked to rotate the shoulder internally and externally, respectively.
2. Pain:

   The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation , and to describe the place and the degree of the pain.
3. Upper limbs function:

   To investigate the motor shoulder function DASH (Disabilities of the Arm, Shoulder and Hand Questionnaire) questionnaire will be used. It assesses the functional capacity in upper limb diseases and measures the skills to do certain activities, as well as the symptoms. It consists of 30 self-administered questions and two optional modules, for sports or musical activities and work activities. The 30 items evaluate the degree of difficulty in the performance of activities; the intensity of the symptoms of pain, weakness, stiffness and numbness; the commitment of social activities; the difficulty to sleep and psychological commitment by reference to the week preceding the instrument application. The final score ranges from zero to one hundred, and the higher the score, the higher the upper limb dysfunction (arm, shoulder or hand).
4. Dehiscence:

   Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution. A Nikon Coolpix S3000 camera will be used.
5. Seroma:

The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer, who will be submitted to breast surgery (radical or conservative), followed by immediate reconstruction: alloplastic (tissue expander or breast implant) or oncoplastic (breast reduction or contralateral symmetrization).

Exclusion Criteria:

* Patients that will be submitted to bilateral oncology surgery, reconstruction with autologous tissue or breast surgery without reconstruction. Patients with motor or neurological deficits prior to surgery, with cognitive impairment and those that do not accept to participate.
* Patients who need to undergo new surgical procedures during the postoperative follow-up period and those who do not appear to postoperative evaluations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 07 days after surgery assessment | One week before surgery on average and 07 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 15 days after surgery assessment | One week before surgery on average and 15 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 30 days after surgery assessment | One week before surgery on average and 30 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 60 days after surgery assessment | One week before surgery on average and 60 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 90 days after surgery assessment | One week before surgery on average and 90 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.
Change in shoulder range of motion from preoperative assessment (one week before surgery on average) at 180 days after surgery assessment | One week before surgery on average and 180 days after surgery
  The shoulder ROM will be assessed with a goniometer for flexion, extension, adduction, abduction, internal rotation and external rotation. The movements will be performed actively.

SECONDARY OUTCOMES:
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 07 days after surgery assessment | One week before surgery on average and 07 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 15 days after surgery assessment | One week before surgery on average and 15 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 30 days after surgery assessment | One week before surgery on average and 30 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 60 days after surgery assessment | One week before surgery on average and 60 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 90 days after surgery assessment | One week before surgery on average and 90 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in self reported pain intensity from preoperative assessment (one week before surgery on average) at 180 days after surgery assessment | One week before surgery on average and 180 days after surgery
  The pain will be evaluated with the Verbal Scale of Pain from zero to ten, where zero is no pain and ten is unbearable pain. The patient will be asked if there is pain at the moment of evaluation, and to describe the place and the degree of the pain.
Change in upper limbs function from preoperative assessment (one week before surgery on average) at 30 days after surgery assessment | One week before surgery on average and 30 days after surgery
  To investigate the motor shoulder function DASH (Disabilities of the Arm, Shoulder and Hand Questionnaire) questionnaire will be used. It assesses the functional capacity in upper limb diseases and measures the skills to do certain activities, as well as the symptoms. It consists of 30 self-administered questions and two optional modules, for sports or musical activities and work activities. The 30 items evaluate the degree of difficulty in the performance of activities; the intensity of the symptoms of pain, weakness, stiffness and numbness; the commitment of social activities; the difficulty to sleep and psychological commitment by reference to the week preceding the instrument application. The final score ranges from zero to one hundred, and the higher the score, the higher the upper limb dysfunction (arm, shoulder or hand).
Change in upper limbs function from preoperative assessment (one week before surgery on average) at 90 days after surgery assessment | One week before surgery on average and 90 days after surgery
  To investigate the motor shoulder function DASH (Disabilities of the Arm, Shoulder and Hand Questionnaire) questionnaire will be used. It assesses the functional capacity in upper limb diseases and measures the skills to do certain activities, as well as the symptoms. It consists of 30 self-administered questions and two optional modules, for sports or musical activities and work activities. The 30 items evaluate the degree of difficulty in the performance of activities; the intensity of the symptoms of pain, weakness, stiffness and numbness; the commitment of social activities; the difficulty to sleep and psychological commitment by reference to the week preceding the instrument application. The final score ranges from zero to one hundred, and the higher the score, the higher the upper limb dysfunction (arm, shoulder or hand).
Dehiscence at 07 days after surgery assessment | 07 days after surgery
  Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution.
Dehiscence at 15 days after surgery assessment | 15 days after surgery
  Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution.
Dehiscence at 30 days after surgery assessment | 30 days after surgery
  Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution.
Dehiscence at 60 days after surgery assessment | 60 days after surgery
  Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution.
Dehiscence at 90 days after surgery assessment | 90 days after surgery
  Dehiscence wil be assessed by inspection and palpation. It will be described "presence" or "absence" of dehiscence and its location. The wound conditions will be described, with observation of necrosis and infection. Signs of infection such as redness, hyperthermia and secretion will be reported. The size of dehiscence will be described: in relation to the amount of opening points, in case of several opened points; or in centimeters (assessed per tape). Photographic record of dehiscence will be done, for better analysis and comparison of evolution.
Seroma at 07 days after surgery assessment | 07 days after surgery
  The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.
Seroma at 15 days after surgery assessment | 15 days after surgery
  The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.
Seroma at 30 days after surgery assessment | 30 days after surgery
  The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.
Seroma at 60 days after surgery assessment | 60 days after surgery
  The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.
Seroma at 90 days after surgery assessment | 90 days after surgery
  The seroma evaluation will be performed by inspection and palpation. There will be description of "presence" or "absence" of seroma, location and the number of punctures made by the medical team and drained quantity, when necessary.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Almeida Rizzi SKL, Haddad CAS, Giron PS, Figueira PVG, Estevao A, Elias S, Nazario ACP, Facina G. Early Free Range-of-Motion Upper Limb Exercises After Mastectomy and Immediate Implant-Based Reconstruction Are Safe and Beneficial: A Randomized Trial. Ann Surg Oncol. 2020 Nov;27(12):4750-4759. doi: 10.1245/s10434-020-08882-z. Epub 2020 Jul 28. PMID 32725529